CLINICAL TRIAL: NCT00903838
Title: A Multicenter, Randomized, Double Blind, Pramipexole Controlled Pilot Study to Assess Efficacy and Safety of Pardoprunox as Adjunct Therapy to L-dopa in the Treatment of Patients With Parkinson's Disease Experiencing Motor Fluctuations and Dyskinesia.
Brief Title: A Pilot Study to Assess Efficacy and Safety of Pardoprunox as Adjunct Therapy to L-dopa in the Treatment of Patients With Parkinson's Disease Experiencing Motor Fluctuations and Dyskinesia.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on 31 May, 2011, due to strategic considerations.
Sponsor: Abbott Products (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S308.2.008; 2008-000400-81 (EudraCT Number)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Advanced Stage Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — pardoprunox; Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: pardoprunox
- 2 (Active Comparator)
  Interventions: Drug: pramipexole

INTERVENTIONS:
Drug: pardoprunox — 1.5 to 12 mg/day
  Arms: 1
Drug: pramipexole — 0.75-4.5 mg/day
  Arms: 2

SUMMARY:
This is a multicenter, randomized, double blind, pramipexole-controlled parallel group study of pardoprunox as adjunctive treatment to levodopa.

DETAILED DESCRIPTION:
Approximately 44 patients are to be randomized in a 3:1 ratio to two possible treatment groups, pardoprunox and pramipexole, respectively. The first part of the study will be blinded and consists of a minimum 1-week screening period, a 4-week switch and stabilization period and an 8-week maintenance period. The second part of the study will be open label pardoprunox treatment with a dose adjustment period of 4 weeks followed by long term maintenance treatment.

ELIGIBILITY:
Inclusion Criteria

* Patients who have signed informed consent
* Diagnosis of idiopathic Parkinson's Disease
* Stable treatment with L-dopa and dopamine agonist for at least 28 days prior to randomization
* Presence of a recognizable ON and OFF state (motor fluctuations)
* Minimum hours of OFF-time per day of 1.5 hours (during waking hours including early morning akinesia) as recorded per baseline diaries
* Minimum hours of ON time with troublesome dyskinesia of 2 hours (during waking hours) as recorded per baseline diaries
* Prevalent expression of severely disabling dyskinesias during the waking day, i.e. dyskinesias are present at least 25% of the waking hours (UPDRS Part 4 item 32 >= 2) in combination with a degree of disability which is moderate or higher (UPDRS Part 4 item 33 >=2)

Exclusion Criteria

* Diagnosis is unclear or a suspicion of other parkinsonian syndromes
* Patients who have undergone surgery for the treatment of PD

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in ON-time without dyskinesia | 16 weeks

SECONDARY OUTCOMES:
Change from baseline in ON-time with (troublesome) dyskinesia; OFF-time; UDysRS, UPDRS (part II + III during ON and OFF state) and Part 4 | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Bronzova, MD, Study Director — Abbott Healthcare Products B.V.
Locations (9):
- Germany (4):
  - Site Reference ID/Investigator# 45433, Göttingen
  - Site Reference ID/Investigator# 45428, Kassel
  - Site Reference ID/Investigator# 45422, Tübingen
  - Site Reference ID/Investigator# 45427, Ulm
- Italy (3):
  - Site Reference ID/Investigator# 45435, Cassino
  - Site Reference ID/Investigator# 45436, Chieti Scalo
  - Site Reference ID/Investigator# 45437, Rome
- Portugal (2):
  - Site Reference ID/Investigator# 45438, Coimbra
  - Site Reference ID/Investigator# 45439, Lisbon